CLINICAL TRIAL: NCT00866281
Title: A Phase I/II, Open-label, Dose-escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Twice Daily Oral Midostaurin and to Evaluate the Preliminary Clinical and Pharmacodynamic Response in Pediatric Patients With Relapsed or Refractory Leukemia
Brief Title: A Study of the Safety and Preliminary Efficacy of Oral Midostaurin (PKC412) in Relapsed or Refractory Pediatric Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Despite considerable efforts to boost recruitment during the final year of the study, no new patients were enrolled.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPKC412A2114; 2008-006931-11 (EudraCT Number)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Acute Myeloid Leukemia; AML; Acute Lymphoblastic Leukemia; ALL; midostaurin; PKC412; Pediatric relapsed or refractory FLT3 positive Acute Myeloid Leukemia; Pediatric relapsed or refractory Mixed-lineage leukemia gene rearranged Acute Lymphoblastic leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — midostaurin

ARMS (2):
- 30 mg/m^2 bid (Experimental): Participants received bodyweight and body surface area (BSA) stratified dose of midostaurin 30 mg/m^2 twice daily (bid) through oral route. The total daily dose in 30 mg/m^2 bid cohort was 60 mg/m^2.
  Interventions: Drug: midostaurin
- 60 mg/m^2 bid (Experimental): Participants received bodyweight and BSA stratified dose of midostaurin 60 mg/m^2 bid through oral route. The total daily dose in 60 mg/m^2 bid cohort was 120 mg/m^2.
  Interventions: Drug: midostaurin

INTERVENTIONS:
Drug: midostaurin — Midostaurin 25 mg/mL oral solution was provided in bottles of 50 mL, administered with water. The pediatric starting dose of midostaurin was set at 30 mg/m2 bid and was not to exceed 60 mg/m2 bid.
  Other Names: PKC412

SUMMARY:
This is a phase I/II pediatric dose-ranging study that will evaluate the safety, tolerability, clinical response, pharmacokinetics and pharmacodynamics of midostaurin in patients <18 years of age who have relapsed or refractory acute leukemias that may benefit from administration of midostaurin, including MLL-rearranged ALL and FLT3 positive AML.

ELIGIBILITY:
Inclusion Criteria:

* Mixed-lineage leukemia (MLL) gene rearranged Acute Lymphoblastic Leukemia (ALL), that does not respond to treatment or has relapsed from prior treatment; or FLT3 mutated Acute Myeloid Leukemia (AML) that does not respond to a second treatment or has relapsed from 2 prior treatments
* Normal organ function, and chest x-ray
* Expected survival greater than 8 weeks
* Can care for most of personal needs and perform at least minimum activity

Exclusion Criteria:

* Patients with symptomatic leukemic central nervous system involvement or isolated extramedullary leukemia
* Patients must not have received other treatments for leukemia within a predefined time period, 72 hours for medications, 2 months for transplants
* Patients with heart function that is not normal
* Patients with HIV or hepatitis
* Patients with another severe disease or medical condition besides leukemia Other protocol-defined inclusion/exclusion criteria may apply

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Seattle Children's Hospital CPKC412A2114, Seattle, Washington, United States
- Novartis Investigative Site, Paris, France
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in 5 countries.
Pre-assignment Details: A total of 22 participants were enrolled in the study.
Groups:
- Cohort 1: Midostaurin (30 Milligrams/Meters^2): Participants received bodyweight and body surface area (BSA) stratified dose of midostaurin 30 mg/m^2 twice daily (bid) through oral route. The total daily dose in 30 mg/m^2 bid cohort was 60 mg/m^2.
- Cohort 2: Midostaurin (60 mg/m^2): Participants received bodyweight and BSA stratified dose of midostaurin 60 mg/m^2 bid through oral route. The total daily dose in 60 mg/m^2 bid cohort was 120 mg/m^2.
Period: Overall Study
Arm/Group | Cohort 1: Midostaurin (30 Milligrams/Meters^2) | Cohort 2: Midostaurin (60 mg/m^2)
Started | 7 | 15
Completed | 0 | 0
Not Completed | 7 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by participants | 3 | 0
Not completed — Disease progression | 3 | 11
Not completed — New cancer therapy | 0 | 4

BASELINE CHARACTERISTICS:
Population: The analysis was performed in full analysis set (FAS) population, defined as all participants to whom study treatment was assigned.
Groups:
- Cohort 1: Midostaurin (30 Milligrams/Meters^2): Participants received body-weight and BSA stratified dose of midostaurin 30 mg/m^2 bid through oral route. The total daily dose in 30 mg/m^2 bid cohort was 60 mg/m^2.
- Cohort 2: Midostaurin (60 mg/m^2): Participants received body-weight and BSA stratified dose of midostaurin 60 mg/m^2 bid through oral route. The total daily dose in 60 mg/m^2 bid cohort was 120 mg/m^2.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Midostaurin (30 Milligrams/Meters^2) | Cohort 2: Midostaurin (60 mg/m^2) | Total
Number analyzed (Participants) | 7 | 15 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.65 (7.479) | 6.50 (6.903) | 7.50 (7.070)
Age, Customized [Number; unit: participants]
  Infants and toddlers (28 days-23 months) | 2 | 9 | 11
  Children (2--11 years) | 1 | 1 | 2
  Adolescents (12--17 years) | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Midostaurin- Posterior Probability of DLT
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced dose limiting toxicity (DLT), based on a Bayesian logistic regression model (BLRM) employing the escalation with overdose control (EWOC) principle. A DLT was defined as a grade 3 or 4 non-hematological adverse event (AE) or abnormal laboratory value related to study drug. Mean and the 95% posterior probability estimates of having a DLT by age strata and dose is presented. Estimation of MTD and/or recommended dose for expansion (RDE) at the dose-escalation phase of the study was based upon the estimation of the probability of DLT for participants in the dose-determining set (DDS).
Time Frame: Baseline, End of dose escalation phase (6 months)
Population: The analysis was performed in dose determining set (DDS) population. Here, 'n' signifies the number of evaluable participants for this measure.
Measure: Mean (97.5% Confidence Interval); unit: probability estimates
Groups:
- Cohort 1: Midostaurin (30 Milligrams/Meters^2): Participants received bodyweight and BSA stratified dose of midostaurin 30 mg/m^2 bid through oral route. The total daily dose in 30 mg/m^2 bid cohort was 60 mg/m^2.
Arm/Group | Cohort 1: Midostaurin (30 Milligrams/Meters^2) | Cohort 2: Midostaurin (60 mg/m^2)
Number analyzed (Participants) | 6 | 11
probability estimates
  Younger stratum (≥ 3months -≤ 2 years): (n=2, 5) | 0.03 [0 to 0.16] | 0.10 [0.01 to 0.33]
  Older stratum (>2 years- <18years): (n=4,6) | 0.03 [0 to 0.13] | 0.08 [0.01 to 0.26]

2. Secondary Outcome: Percentage of Participants With Best Overall Response by Indication
Description: The best overall clinical response was determined as per the clinical assessment done by the investigator. Responders were defined as all participants with a best clinical response of leukemia free state, morphological complete remission, incomplete morphological complete remission, partial remission, bone marrow blast response, bone marrow minor blast response, peripheral blood blast response, minor peripheral blood blast response. Participants with stable disease, progressive disease and with missing tumour assessment or who discontinued the study or who died before having their first assessment were considered as non-responders. Stable disease was defined as failure to achieve any of the above response. Progressive disease was defined as doubling of the bone marrow blast percentage from baseline in participants with <40% bone marrow blasts at baseline, or a 50% increase in bone marrow blast percentage from baseline in participants with >40% bone marrow blasts at baseline,
Time Frame: Baseline, Day 15 (Day 1 of Cycle 2), Day 22 (Day 8 of Cycle 2), Day 29(Day 1 of Cycle 9), End of treatment (up to 24 months after last dose or until death whichever occurred first)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Groups:
- AML Subjects: Subjects with acute myeloid leukemia (AML) and received body-weight stratified dosage midostaurin 30 or 60 mg/m^2.
- MLLr-ALL Subjects: Subjects with mixed lineage leukemia gene- rearranged acute lymphoblastic leukemia (MLLr-ALL) and received body-weight stratified dosage midostaurin 30 or 60 mg/m^2.
Arm/Group | AML Subjects | MLLr-ALL Subjects
Number analyzed (Participants) | 9 | 13
Percentage of Participants
  Leukemia free state | 0 | 0
  Morphological complete remission | 0 | 0
  Incomplete morphological complete remission | 11.1 | 0
  Partial remission | 0 | 0
  Bone marrow blast response | 22.2 | 0
  Bone marrow minor blast response | 0 | 0
  Peripheral blood blast response | 11.1 | 23.1
  Minor peripheral blood blast response | 11.1 | 0
  Stable disease | 44.4 | 7.7
  Progressive disease | 0 | 61.5
  Not Done | 0 | 7.7
  Participants with response | 55.6 | 23.1

3. Secondary Outcome: Time to Response With Midostaurin
Description: Time to response was defined as the time from the date of start of midostaurin treatment to the date of first response. The best overall clinical response was determined as per the clinical assessment done by the investigator. Responders were defined as all participants with a best clinical response of leukemia free state, morphological complete remission, incomplete morphological complete remission, partial remission, bone marrow blast response, bone marrow minor blast response, peripheral blood blast response, minor peripheral blood blast response. Time to response was calculated by using the formula = (date of first response -date of start of midostaurin) +1 day.
Time Frame: Baseline, End of treatment (up to 24 months after last dose or until death whichever occurred first)
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies number of responders at specified time points for each arm, respectively.
Measure: Median (Full Range); unit: Days
Arm/Group | AML Subjects | MLLr-ALL Subjects
Number analyzed (Participants) | 5 | 3
Days | 14.0 [8.0 to 22.0] | 8.0 [3.0 to 8.0]

4. Secondary Outcome: Overall Survival With Midostaurin
Description: Overall survival (OS) was defined as the time from start of treatment to date of death due to any cause. The percentage (%) event-free probability estimates were obtained from the Kaplan-Meier survival estimates.
Time Frame: Baseline, End of treatment (up to 24 months after last dose or until death whichever occurred first)
Population: The analysis was performed in FAS population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AML Subjects | MLLr-ALL Subjects
Number analyzed (Participants) | 9 | 13
Months | 3.68 [2.727 to 8.312] | 1.35 [0.953 to 2.924]

5. Secondary Outcome: Plasma Concentrations of Midostaurin and Its Metabolites CGP52421 and CGP62221
Description: The plasma concentrations of midostaurin (PKC412) and its two major metabolites, CGP62221 and CGP52421 were determined by using a validated liquid chromatography/tandem mass spectrometry method.
Time Frame: Day 1, Day 5, Day 7, Day 15 (Day 1 of Cycle 2), Day 29 (Day 1 of Cycle 3)
Population: The analysis was performed in pharmacokinetic (PK) set population defined as all safety set participants who had at least one valid (measurable) PK sample of midostaurin, and who had no significant restricted co-medications.
Measure: Mean (Standard Deviation); unit: nanograms/milliliters (ng/mL)
Groups:
- Cohort 1: Midostaurin (30 Milligrams/Meters^2): Participants received bodyweight and body surface area (BSA) stratified dose of midostaurin 30 mg/m^2 bid through oral route. The total daily dose in 30 mg/m^2 bid cohort was 60 mg/m^2.
Arm/Group | Cohort 1: Midostaurin (30 Milligrams/Meters^2) | Cohort 2: Midostaurin (60 mg/m^2)
Number analyzed (Participants) | 7 | 15
nanograms/milliliters (ng/mL)
  PKC412-Cycle 1/Day 1 (1 hour) | 1678 (652.817) | 2330.88 (1290.136)
  PKC412-Cycle 1/Day 1 (2 hour) | 1762.5 (226.771) | 2449.09 (936.039)
  PKC412-Cycle 1/Day 1 (3 hour) | 1891.67 (505.941) | 2287.5 (1421.365)
  PKC412-Cycle 1/Day 1 (12 hour) | 939.17 (347.925) | 2068.85 (2183.946)
  PKC412-Cycle 1/Day 5 (0 hour) | 2444 (936.659) | 2610.1 (2480.716)
  PKC412-Cycle 1/Day 7 (0 hour) | 1945 (643.467) | 2028 (2071.949)
  PKC412-Cycle 2/Day 1 (0 hour) | 1832.5 (773.881) | 726 (379.953)
  PKC412-Cycle 3/Day 1 (0 hour) | 962 (505.146) | 674 (340.776)
  CGP62221-Cycle 1/Day 1 (1 hour) | 106.18 (89.473) | 228.33 (148.469)
  CGP62221-Cycle 1/Day 1 (2 hour) | 208.95 (183.22) | 458.75 (281.882)
  CGP62221-Cycle 1/Day 1 (3 hour) | 333.4 (227.863) | 563.63 (276.938)
  CGP62221-Cycle 1/Day 1 (12 hour) | 424.35 (299.416) | 730.31 (385.698)
  CGP62221-Cycle 1/Day 5 (0 hour) | 3182 (1756.778) | 3360.3 (2002.498)
  CGP62221-Cycle 1/Day 7 (0 hour) | 3390 (1400.071) | 2895 (1893.347)
  CGP62221-Cycle 2/Day 1 (0 hour) | 2380 (728.331) | 1614.14 (1057.585)
  CGP62221-Cycle 3/Day 1 (0 hour) | 1140.67 (189.16) | 1759.2 (923.668)
  CGP52421-Cycle 1/Day 1 (1 hour) | 71.64 (42.325) | 111.58 (78.187)
  CGP52421-Cycle 1/Day 1 (2 hour) | 113.23 (54.831) | 189.65 (128.879)
  CGP52421-Cycle 1/Day 1 (3 hour) | 152.18 (78.405) | 236.19 (144.723)
  CGP52421-Cycle 1/Day 1 (12 hour) | 139.27 (68.198) | 259.52 (148.943)
  CGP52421-Cycle 1/Day 5 (0 hour) | 1018 (259.014) | 1581 (509.208)
  CGP52421-Cycle 1/Day 7 (0 hour) | 1269 (453.963) | 2129 (341.97)
  CGP52421-Cycle 2/Day 1 (0 hour) | 2350 (1110.465) | 2640 (541.018)
  CGP52421-Cycle 3/Day 1 (0 hour) | 2386.67 (277.909) | 3488 (1511.529)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment Related AEs or SAEs and Death During the Study
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes. Treatment related AEs or SAEs were defined as AEs or SAEs that were suspected to be related to study treatment as per investigator. On treatment death was a fatal event leading to permanent cessations of all vital functions of the body.
Time Frame: Baseline (start of study treatment) up to End of treatment (up to 24 months after last dose or until death whichever occurred first)
Population: The analysis was performed in safety set population, defined as the participants who received at least one dose of midostaurin.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: Midostaurin (30 Milligrams/Meters^2) | Cohort 2: Midostaurin (60 mg/m^2)
Number analyzed (Participants) | 7 | 15
Participants
  AEs | 6 | 15
  AEs suspected to be drug related | 1 | 2
  On-treatment death | 2 | 3
  SAEs | 3 | 6
  SAEs suspected to be drug related | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious Adverse Events are monitored from date of First Participant First Visit (FPFV) up to Last Participant Last Visit (LPLV), 24 weeks and all other adverse events are monitored from First Participant First Treatment (FPFT) up to LPLV, 20 weeks
Arm/Group | Cohort 1: Midostaurin (30 Milligrams/Meters^2) | Cohort 2: Midostaurin (60 mg/m^2)
Serious Adverse Events (participants affected / at risk) | 3/7 | 6/15
Other Adverse Events (participants affected / at risk) | 6/7 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Midostaurin (30 Milligrams/Meters^2) (N=7) | Cohort 2: Midostaurin (60 mg/m^2) (N=15)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Tongue Oedema (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Tongue Injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Blast Cell Count Increased (Investigations) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Midostaurin (30 Milligrams/Meters^2) (N=7) | Cohort 2: Midostaurin (60 mg/m^2) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 9
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 7
Oral Mucosal Exfoliation (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Oral Pruritus (Gastrointestinal disorders) | 0 | 1
Tongue Discolouration (Gastrointestinal disorders) | 0 | 1
Tooth Loss (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 12
Asthenia (General disorders) | 0 | 1
Catheter Site Inflammation (General disorders) | 0 | 1
Catheter Site Pain (General disorders) | 0 | 1
Crying (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Feeling Abnormal (General disorders) | 0 | 1
Generalised Oedema (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 7
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1
Enterobacter Infection (Infections and infestations) | 1 | 0
Enterobacter Sepsis (Infections and infestations) | 1 | 0
Febrile Infection (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 4
Aspartate Aminotransferase Increased (Investigations) | 1 | 4
Blood Albumin Decreased (Investigations) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Blood Fibrinogen Decreased (Investigations) | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1
Blood Phosphorus Decreased (Investigations) | 0 | 1
Cardiac Murmur (Investigations) | 0 | 1
Electrocardiogram Qt Prolonged (Investigations) | 0 | 2
Haemoglobin Decreased (Investigations) | 0 | 1
Heart Sounds Abnormal (Investigations) | 0 | 1
Lipase Increased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 2
Weight Increased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 2
White Blood Cell Count Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 4
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 5
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Mood Altered (Psychiatric disorders) | 0 | 3
Nightmare (Psychiatric disorders) | 0 | 1
Breast Haematoma (Reproductive system and breast disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1
Capillary Leak Syndrome (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early since despite considerable efforts to boost recruitment, no new participants were enrolled in the final year of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e, data from all sites) in the clinical trial.